CLINICAL TRIAL: NCT02748018
Title: Multi-center, Randomized, Parallel, Adaptive, Controlled Trial in Adult and Pediatric Patients With Type 1 Diabetes Using Hybrid Closed Loop System and Control (CSII, MDI and SAP) at Home
Brief Title: Multi-center Trial in Adult and Pediatric Patients With Type 1 Diabetes Using Hybrid Closed Loop System and Control at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP 304
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: There will be three cohorts sequentially enrolled for the study. Cohort 1: Continuous Subcutaneous Insulin Infusion (CSII cohort): randomized to HCL (treatment arm) or CSII (Control arm) Cohort 2: Multiple Daily Injections (MDI cohort): randomized to HCL (treatment arm) or MDI (Control arm) Cohort 3: Sensor-Augmented Pump therapy (SAP cohort): randomized to HCL (treatment arm) or SAP (Control arm) Note: Subjects 2-6 years of age will automatically enter the HCL arm at the end of the run-in period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Hybrid Closed Loop Arm (Experimental): The HCL Arm will use the MiniMed System (i.e., using Auto Mode) for 6 months during the study period.
  Interventions: Device: 670G and 770G Insulin Pump
- Control Arm (Active Comparator): The Control Arm will use individual subject's current diabetes therapy: CSII (Continuous Subcutaneous Insulin Infusion), MDI (Multiple Daily Injections) or SAP (Sensor Augmented Pump). Each cohort (CSII, MDI, or SAP) will be used as the control arm to be compared to the experimental arm (HCL).
  Interventions: Device: Subject's Current Diabetes Therapy

INTERVENTIONS:
Device: 670G and 770G Insulin Pump — Medtronic 670G and 770G Hybrid Closed Loop Systems
  Arms: Hybrid Closed Loop Arm
Device: Subject's Current Diabetes Therapy — Subject will use current diabetes therapy: CSII (Continuous Subcutaneous Insulin Infusion), MDI (Multiple Daily Injections) or SAP (Sensor Augmented Pump).
  Arms: Control Arm

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Hybrid Closed Loop system (HCL) in adult and pediatric patients with type 1 diabetes in the home setting. A diverse population of patients with type 1 diabetes will be studied. The study population will have a large range for duration of diabetes and glycemic control, as measured by glycosylated hemoglobin (A1C). They will be enrolled in the study regardless of their prior diabetes regimen, including using Multiple Daily Injections (MDI), Continuous Subcutaneous Insulin Infusion (CSII) or Sensor-Augmented Pump therapy (SAP)

DETAILED DESCRIPTION:
This is a 6 month, multi-center, randomized, parallel, adaptive study in type 1 diabetes with a 6 month continuation period. The study will have three periods, per Cohort:

1. Run-in Period: The run-in period can be up to 60 days during which time a blinded CGM sensor will be worn for two weeks.
2. Study Period: There will be a 6 month randomized study period with two arms: The HCL system and Control. The primary and secondary endpoints will be evaluated during this period only.
3. Continuation Period: There will be a 6 month continuation period during which time all subjects will use the HCL system with Auto Mode. Only the safety endpoint will be evaluated during this period.

Up to 1500 subjects will be enrolled in order to have 1000 subjects complete the study. Up to 70 investigational Centers in the US, Europe, Canada, Australia and New Zealand will be enrolled.

ELIGIBILITY:
Inclusion Criteria

1. Subject is age 2-80 years at time of screening

   1. US, Canada, Australia and New Zealand: Subjects 2-80 years of age will be allowed to enroll in the post approval study.
   2. Europe: Only subjects ≥7 years of age are allowed to enroll in the post-market study.
2. Subjects who are 2-21 years are determined by the investigator to have the appropriate, requisite support (family, caregiver or social network) to successfully participate in this study
3. Subject must have a minimum daily insulin requirement (Total Daily Dose) of equal to or greater than 8 units/day
4. Subjects who are determined by the investigator to be psychologically sound in order to successfully participate in this study
5. Subject has been diagnosed with type 1 diabetes for at least three months Note: Determination of classification for diabetes will be based on American Diabetes Association Clinical Practice Guidelines accounting for several patient characteristics such as: age of onset, patient's weight or BMI, history of diabetic ketoacidosis, history of therapy management, if available in the medical records.
6. Subject must be on one of the following management therapies:

   1. Multiple daily injections defined by use of rapid analogue with meals and approved long acting analogue (e.g. detemir or glargine) with or without CGM
   2. Insulin pump therapy with or without CGM
7. Subject is willing to perform ≥ 4 finger stick blood glucose measurements daily
8. Subject is willing to perform required study procedures
9. Subject is willing to wear the system continuously throughout the study for at least 80% of the time.
10. Subject is willing to upload data at least weekly from the study pump/meter, must have Internet access and a computer system that meets the requirements for uploading the study pump/meter for data collection
11. Subject must be willing to use the study glucose meter system (i.e. along with study meter strips).
12. If subject has celiac disease, it has been adequately treated as determined by the investigator
13. Subject with the diagnosis of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease, within 1 year of screening, will be included in the study with the consent of the Investigator
14. Subject is willing to take one of the following insulins and can financially afford to use either of the 2 insulin preparations throughout the course of the study (i.e. co-payments for insulin with insurance or able to pay full amount)

    1. Humalog® (insulin lispro injection)
    2. NovoLog® (insulin aspart)

Exclusion Criteria:

1. Subject participated in any Closed Loop study in the past.
2. Subject is unable to tolerate tape adhesive in the area of sensor placement
3. Subject has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, rash, Staphylococcus infection) or area of infusion set placement
4. Women of child-bearing potential who have a positive pregnancy test at screening or plan to become pregnant during the course of the study
5. Subject is being treated for hyperthyroidism at time of screening
6. Subject has an abnormality (out of reference range) in thyroid-stimulating hormone (TSH) at time of screening visit. TSH is not required for subjects 2-13 years of age.
7. Subject has taken any oral, injectable, or IV glucocorticoids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study.
8. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks
9. Subject is currently abusing illicit drugs or marijuana
10. Subject is currently abusing prescription drugs
11. Subject is currently abusing alcohol
12. Subject is using pramlintide (Symlin), SGLT2 inhibitors, GLP agonists, biguanides, DPP-4 inhibitors or sulfonylureas at time of screening
13. Subject is using hydroxyurea at the time of screening or plans to use it during the study
14. Subject has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator
15. Subject has a sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
16. Subject plans to receive red blood cell transfusion or erythropoietin over the course of study participation
17. Subject diagnosed with current moderate to severe eating disorder such as anorexia or bulimia
18. Subject has been diagnosed with chronic kidney disease requiring dialysis or resulting in chronic anemia
19. Subjects who are currently being actively treated for cancer.
20. Subject who is designated as a research staff member for this study

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 959 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (25):
  - Scripps Health System, La Jolla, California
  - Stanford University, Palo Alto, California
  - Center of Excellence in Diabetes & Endocrinology, Sacramento, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - SoCal Diabetes, Torrance, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center, Aurora, Colorado
  - University of South Florida Diabetes Center, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Rocky Mountain Diabetes, Idaho Falls, Idaho
  - Indiana University Health Riley Hospital for Children, Indianapolis, Indiana
  - IDERC, Des Moines, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Grunberger Diabetes Institute, Bloomfield Hills, Michigan
  - Initernational Diabetes Center, Minneapolis, Minnesota
  - International Diabetes Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University St. Louis, St Louis, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - Sanford Health, Sioux Falls, South Dakota
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Diabetes and Glandular Disease Clinic, P.A., San Antonio, Texas
  - Rainier Clinical Research, Renton, Washington
  - University of Washington, Seattle, Washington
- Canada (2):
  - Westminster Endocrine & Diabetes Research Society, New Westminster, British Columbia
  - Children's Hospital of Eastern Ontario, Ottawa
- France (2):
  - Hôpital Necker Enfants Malades, Paris
  - HCL - Lyon Sud, Pierre-Bénite
- Diabeteszentrum für Kinder und Jugendliche, Kinder- und Jugendkrankenhaus Auf der Bult, Hanover, Germany
- A.S.S.T. Spedali Civili, Brescia, Italy
- New Zealand (2):
  - New Zealand Clinical Research, Christchurch
  - Dunedin Public Hospital, Dunedin
- Hospital Universitario Virgen del Rocío, Seville, Spain
- Dept Internal Medicine, Örebro University Hospital, Örebro, Sweden
- Cambridge University Hospitals NHS Foundation Trust - Addenbrooke's Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jendle JH, Garg SK, Thivolet C, Weinstock RS, Hirsch IB, Evans M, Griffin KJ, Philis-Tsimikas A, Wheeler BJ, Kipnes MS, Carlson AL, Buckingham BA, Bhargava A, Bode BW, Lawson ML, Criego AB, McGill JB, Reed JCH, Prakasam G, Grunberger G, Girelli A, Martinez-Brocca MA, Christiansen MP, de Bock MI, Kudva YC, Lee SW, Yovanovich C, Shin JJ, Cordero TL, McVean JJF, Vigersky RA. Automated basal insulin delivery versus multiple daily injections in type 1 diabetes: results from a randomized parallel controlled trial. Front Endocrinol (Lausanne). 2025 Dec 19;16:1716587. doi: 10.3389/fendo.2025.1716587. eCollection 2025. PMID 41488135

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first subject enrollment: 25MAY2017, Date of last subject visit (of study period): 09MAY2023 Date of last subject visit (of continuation period): 01NOV2023
Pre-assignment Details: 870 (298 in CSII Cohort, 248 in MDI Cohort, 324 in SAP Cohort) subjects entered the study period.
Groups:
- CSII Cohort: Treatment Arm: In the run-in period, subjects were on CSII. In the study period, subjects started using the MiniMed system (i.e., using Auto Mode). In the continuation period, all subjects were using the Hybrid Closed Loop system.
- CSII Cohort: Control Arm: In the run-in period, subjects were on CSII. In the study period, subjects used the MiniMed pump without CGM. In the continuation period, all subjects were using the Hybrid Closed Loop system.
- MDI Cohort: Treatment Arm: In the run-in period, subjects were on MDI. In the study period, subjects started using the MiniMed system (i.e., using Auto Mode). In the continuation period, all subjects were using the Hybrid Closed Loop system.
- MDI Cohort: Control Arm: In the run-in period, subjects were on MDI. In the study period, subjects continued to use MDI. In the continuation period, all subjects were using the Hybrid Closed Loop system.
- SAP Cohort: Treatment Arm: In the run-in period, subjects were on SAP. In the study period, subjects started using the MiniMed system (i.e., using Auto Mode). In the continuation period, all subjects were using the Hybrid Closed Loop system.
- SAP Cohort: Control Arm: In the run-in period, subjects were on SAP. In the study period, subjects continued to use SAP therapy using the MiniMed system (SAP without Low Management Suspend on Low, Low Management Suspend before low or Auto Mode). In the continuation period, all subjects were using the Hybrid Closed Loop system.
Period: Study Period
Arm/Group | CSII Cohort: Treatment Arm | CSII Cohort: Control Arm | MDI Cohort: Treatment Arm | MDI Cohort: Control Arm | SAP Cohort: Treatment Arm | SAP Cohort: Control Arm
Started (Subjects entering the study period (randomized)) | 150 | 148 | 126 | 122 | 164 | 160
Completed | 140 | 138 | 117 | 109 | 146 | 146
Not Completed | 10 | 10 | 9 | 13 | 18 | 14
Not completed — Adverse Event | 1 | 3 | 4 | 0 | 3 | 3
Not completed — Withdrawal by Subject | 7 | 4 | 4 | 11 | 12 | 10
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 2 | 2 | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 1
Period: Continuation Period
Arm/Group | CSII Cohort: Treatment Arm | CSII Cohort: Control Arm | MDI Cohort: Treatment Arm | MDI Cohort: Control Arm | SAP Cohort: Treatment Arm | SAP Cohort: Control Arm
Started | 140 | 138 | 117 | 109 | 146 | 146
Completed | 134 | 127 | 110 | 99 | 131 | 140
Not Completed | 6 | 11 | 7 | 10 | 15 | 6
Not completed — Adverse Event | 2 | 0 | 1 | 1 | 1 | 4
Not completed — Withdrawal by Subject | 3 | 5 | 3 | 9 | 11 | 1
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 1 | 0
Not completed — Pregnancy | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 2 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Subjects Entered the Study Period
Groups:
- Total: Total of all reporting groups
Arm/Group | CSII Cohort: Treatment Arm | CSII Cohort: Control Arm | MDI Cohort: Treatment Arm | MDI Cohort: Control Arm | SAP Cohort: Treatment Arm | SAP Cohort: Control Arm | Total
Number analyzed (Participants) | 150 | 148 | 126 | 122 | 164 | 160 | 870
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.0 (19.8) | 35.1 (18.1) | 33.6 (19.6) | 37.9 (19.2) | 36.4 (21.3) | 39.2 (21.4) | 37.1 (20.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 90 | 38 | 42 | 90 | 83 | 414
  Male | 79 | 58 | 88 | 80 | 74 | 77 | 456
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 6 | 16 | 7 | 4 | 45
  Not Hispanic or Latino | 141 | 144 | 109 | 95 | 154 | 156 | 799
  Unknown or Not Reported | 1 | 0 | 11 | 11 | 3 | 0 | 26

OUTCOME MEASURES:

1. Primary Outcome: CSII Cohort: Baseline A1C > 8%: Change in A1C (∆A1C)
Description: CSII Cohort: Change in A1C from baseline to the end of the six-month treatment period, defined as A1C measured at the six-month treatment visit minus A1C measured at the randomization visit, for subjects with baseline A1C > 8%
Time Frame: Baseline and end of 6-month study period
Population: Study period: 298 subjects in CSII cohort. 147 subjects have available measurements in the baseline A1C > 8% group.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | CSII Cohort: Treatment Arm | CSII Cohort: Control Arm
Number analyzed (Participants) | 74 | 73
Percentage of HbA1c | -1.6 (1.3) | -0.8 (0.9)
Statistical Analysis 1: Comparison: CSII Cohort: Treatment Arm vs CSII Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Change in A1C with Multiple Imputation; Mean Difference (Final Values) = -0.8, 97.5% CI 1-sided [upper limit -0.4]

2. Primary Outcome: CSII Cohort: Baseline A1C ≤ 8%: Time in Hypoglycemic Range
Description: CSII Cohort: Time with sensor glucose (SG) below 70 mg/dL (3.9mmol/L) during the six-month study period, for subjects with baseline A1c ≤ 8%
Time Frame: 6 months study period
Population: Study period: 298 subjects in CSII cohort. 129 subjects have available measurements in the baseline A1C ≤ 8% group.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | CSII Cohort: Treatment Arm | CSII Cohort: Control Arm
Number analyzed (Participants) | 66 | 63
Percentage of Time | 2.4 (1.9) | 7.3 (5.3)
Statistical Analysis 1: Comparison: CSII Cohort: Treatment Arm vs CSII Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Hypoglycemic Range (%); Mean Difference (Final Values) = -4.9, 97.5% CI 1-sided [upper limit -3.6]

3. Primary Outcome: MDI Cohort: Baseline A1C > 8%: Change of A1C (∆A1C)
Description: MDI Cohort: Change in A1C from baseline to the end of the six-month treatment period, defined as A1C measured at the six-month treatment visit minus A1C measured at the randomization visit, for subjects with baseline A1c > 8%
Time Frame: Baseline and end of 6-month study period
Population: Study period: 248 subjects in MDI cohort. 94 subjects have available measurements in the baseline A1C > 8% group.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | MDI Cohort: Treatment Arm | MDI Cohort: Control Arm
Number analyzed (Participants) | 50 | 44
Percentage of HbA1c | -1.4 (1.1) | -0.6 (0.9)
Statistical Analysis 1: Comparison: MDI Cohort: Treatment Arm vs MDI Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Change in A1C with Multiple Imputation; Mean Difference (Final Values) = -0.7, 97.5% CI 1-sided [upper limit -0.3]

4. Primary Outcome: MDI Cohort: Baseline A1C ≤ 8%: Time in Hypoglycemic Range
Description: MDI Cohort: Time with sensor glucose (SG) below 70 mg/dL (3.9mmol/L) during the six-month study period, for subjects with baseline A1c ≤ 8%
Time Frame: 6 months study period
Population: Study period: 248 subjects in MDI cohort. 120 subjects have available measurements in the baseline A1C ≤ 8% group.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | MDI Cohort: Treatment Arm | MDI Cohort: Control Arm
Number analyzed (Participants) | 65 | 55
Percentage of Time | 2.8 (2.7) | 7.5 (6.1)
Statistical Analysis 1: Comparison: MDI Cohort: Treatment Arm vs MDI Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Hypoglycemic Range (%); Mean Difference (Final Values) = -4.8, 97.5% CI 1-sided [upper limit -3.1]

5. Primary Outcome: SAP Cohort: Baseline A1C > 8%: Change of A1C (∆A1C)
Description: SAP Cohort: Change in A1C from baseline to the end of the six-month treatment period, defined as A1C measured at the six-month treatment visit minus A1C measured at the randomization visit, for subjects with baseline A1c > 8%
Time Frame: Baseline and end of 6-month study period
Population: Study period: 324 subjects in SAP cohort. 108 subjects have available measurements in the baseline A1C > 8% group.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | SAP Cohort: Treatment Arm | SAP Cohort: Control Arm
Number analyzed (Participants) | 54 | 54
Percentage of HbA1c | -0.6 (0.8) | -0.6 (1.0)
Statistical Analysis 1: Comparison: SAP Cohort: Treatment Arm vs SAP Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Change in A1C with Multiple Imputation; Mean Difference (Final Values) = 0.0, 97.5% CI 1-sided [upper limit 0.3]

6. Primary Outcome: SAP Cohort: Baseline A1C ≤ 8%: Time in Hypoglycemic Range
Description: SAP Cohort: Time with sensor glucose (SG) below 70 mg/dL (3.9mmol/L) during the six-month study period, for subjects with baseline A1c ≤ 8%
Time Frame: 6 months study period
Population: Study period: 324 subjects in SAP cohort. 177 subjects have available measurements in the baseline A1c ≤ 8% group.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | SAP Cohort: Treatment Arm | SAP Cohort: Control Arm
Number analyzed (Participants) | 89 | 88
Percentage of Time | 2.5 (2.3) | 3.5 (3.0)
Statistical Analysis 1: Comparison: SAP Cohort: Treatment Arm vs SAP Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Hypoglycemic Range (%); Mean Difference (Final Values) = -1.0, 97.5% CI 1-sided [upper limit -0.2]

7. Secondary Outcome: CSII Cohort: Baseline A1C > 8%: Time in Hypoglycemic Range
Description: CSII Cohort: Time with sensor glucose (SG) below 70 mg/dL (3.9mmol/L) during the six-month study period, for subjects with baseline A1c > 8%
Time Frame: 6 months study period
Population: Study period: 298 subjects in CSII cohort. 136 subjects have available measurements in the baseline A1c > 8% group.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | CSII Cohort: Treatment Arm | CSII Cohort: Control Arm
Number analyzed (Participants) | 74 | 62
Percentage of Time | 2.3 (2.3) | 4.6 (5.2)
Statistical Analysis 1: Comparison: CSII Cohort: Treatment Arm vs CSII Cohort: Control Arm; Test type: Non-Inferiority — Non-inferiority margin: 2%. Test of Treatment Effect on Time in Hypoglycemic Range (%); Mean Difference (Final Values) = -2.2, 97.5% CI 1-sided [upper limit -0.9]

8. Secondary Outcome: CSII Cohort: Baseline A1C ≤ 8%: Change in A1C (∆A1C)
Description: CSII Cohort: Change in A1C from baseline to the end of the six-month treatment period, defined as A1C measured at the six-month treatment visit minus A1C measured at the randomization visit, for subjects with baseline A1c ≤ 8%
Time Frame: Baseline and end of 6-month study period
Population: Study period: 298 subjects in CSII cohort. 131 subjects have available measurements in the baseline A1c ≤ 8% group.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | CSII Cohort: Treatment Arm | CSII Cohort: Control Arm
Number analyzed (Participants) | 66 | 65
Percentage of HbA1c | -0.4 (0.5) | -0.0 (0.6)
Statistical Analysis 1: Comparison: CSII Cohort: Treatment Arm vs CSII Cohort: Control Arm; Test type: Non-Inferiority — Non-inferiority margin: 0.4%. Treatment Effect on Change in A1C with Multiple Imputation; Mean Difference (Final Values) = -0.3, 97.5% CI 1-sided [upper limit -0.1]

9. Secondary Outcome: CSII Cohort: Time in Hypoglycemic Range During Night for All Subjects
Description: CSII Cohort: Time with SG below 70 mg/dL (3.9mmol/L) during Night for all subjects
Time Frame: 6 months study period
Population: Study period: 298 subjects in CSII cohort. 264 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | CSII Cohort: Treatment Arm | CSII Cohort: Control Arm
Number analyzed (Participants) | 140 | 124
Percentage of Time | 2.3 (3.3) | 7.7 (9.4)
Statistical Analysis 1: Comparison: CSII Cohort: Treatment Arm vs CSII Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Hypoglycemic Range (%) During Night; Mean Difference (Final Values) = -5.4, 97.5% CI 1-sided [upper limit -3.7]

10. Secondary Outcome: CSII Cohort: Time in Target Range 70mg/dL (3.9mmol/L) - 180 mg/dL (10.0mmol/L) During Night for All Subjects
Description: CSII Cohort: Time in target range measures the time with SG in target range 70mg/dL (3.9mmol/L) - 180 mg/dL (10.0mmol/L) during Night for all subjects
Time Frame: 6 months study period
Population: Study period: 298 subjects in CSII cohort. 264 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | CSII Cohort: Treatment Arm | CSII Cohort: Control Arm
Number analyzed (Participants) | 140 | 124
Percentage of Time | 73.8 (14.3) | 55.0 (20.8)
Statistical Analysis 1: Comparison: CSII Cohort: Treatment Arm vs CSII Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Target Range (%) During Night; Mean Difference (Final Values) = 18.8, 97.5% CI 1-sided [lower limit 14.5]

11. Secondary Outcome: CSII Cohort: Time in Target Range 70mg/dL (3.9mmol/L) - 180 mg/dL (10.0mmol/L) During Day and Night for All Subjects
Description: CSII Cohort: Time in target range measures the time with SG in target range 70mg/dL (3.9mmol/L) - 180 mg/dL (10.0mmol/L) during Day and Night for all subjects
Time Frame: 6 months study period
Population: Study period: 298 subjects in CSII cohort. 265 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | CSII Cohort: Treatment Arm | CSII Cohort: Control Arm
Number analyzed (Participants) | 140 | 125
Percentage of Time | 67.4 (10.8) | 55.4 (15.0)
Statistical Analysis 1: Comparison: CSII Cohort: Treatment Arm vs CSII Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Target Range (%); Mean Difference (Final Values) = 12.0, 97.5% CI 1-sided [lower limit 8.8]

12. Secondary Outcome: CSII Cohort: Time in Hypoglycemic Range During Day and Night for All Subjects
Description: CSII Cohort: Time with SG below 70 mg/dL (3.9mmol/L) during Day and Night for all subjects
Time Frame: 6 months study period
Population: Study period: 298 subjects in CSII cohort. 265 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | CSII Cohort: Treatment Arm | CSII Cohort: Control Arm
Number analyzed (Participants) | 140 | 125
Percentage of Time | 2.4 (2.1) | 6.0 (5.4)
Statistical Analysis 1: Comparison: CSII Cohort: Treatment Arm vs CSII Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Hypoglycemic Range (%); Mean Difference (Final Values) = -3.6, 97.5% CI 1-sided [upper limit -2.6]

13. Secondary Outcome: CSII Cohort: Change in A1C for All Subjects
Description: CSII Cohort: Change in A1C from baseline to the end of the six-month treatment period, defined as A1C measured at the six-month treatment visit minus A1C measured at the randomization visit for all subjects
Time Frame: Baseline and end of 6-month study period
Population: Study period: 298 subjects in CSII cohort. 278 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | CSII Cohort: Treatment Arm | CSII Cohort: Control Arm
Number analyzed (Participants) | 140 | 138
Percentage of HbA1c | -1.0 (1.2) | -0.4 (0.9)
Statistical Analysis 1: Comparison: CSII Cohort: Treatment Arm vs CSII Cohort: Control Arm; Test type: Superiority — Treatment Effect on Change in A1C with Multiple Imputation; Mean Difference (Final Values) = -0.6, 97.5% CI 1-sided [upper limit -0.3]

14. Secondary Outcome: MDI Cohort: Baseline A1C > 8%: Time in Hypoglycemic Range
Description: MDI Cohort: Time with sensor glucose (SG) below 70 mg/dL (3.9mmol/L) during the six-month study period, for subjects with baseline A1c > 8%
Time Frame: 6 months study period
Population: Study period: 248 subjects in MDI cohort. 88 subjects have available measurements in the baseline A1C > 8% group.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | MDI Cohort: Treatment Arm | MDI Cohort: Control Arm
Number analyzed (Participants) | 50 | 38
Percentage of Time | 1.9 (1.6) | 5.5 (5.9)
Statistical Analysis 1: Comparison: MDI Cohort: Treatment Arm vs MDI Cohort: Control Arm; Test type: Non-Inferiority — Non-inferiority margin: 2%. Test of Treatment Effect on Time in Hypoglycemic Range (%); Mean Difference (Final Values) = -3.6, 97.5% CI 1-sided [upper limit -1.9]

15. Secondary Outcome: MDI Cohort: Baseline A1C ≤ 8%: Change in A1C (∆A1C)
Description: MDI Cohort: Change in A1C from baseline to the end of the six-month treatment period, defined as A1C measured at the six-month treatment visit minus A1C measured at the randomization visit, for subjects with baseline A1c ≤ 8%
Time Frame: Baseline and end of 6-month study period
Population: Study period: 248 subjects in MDI cohort. 130 subjects have available measurements in the baseline A1C ≤ 8% group.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | MDI Cohort: Treatment Arm | MDI Cohort: Control Arm
Number analyzed (Participants) | 65 | 65
Percentage of HbA1c | 0.0 (0.6) | -0.1 (0.5)
Statistical Analysis 1: Comparison: MDI Cohort: Treatment Arm vs MDI Cohort: Control Arm; Test type: Non-Inferiority — Non-inferiority margin: 0.4%. Treatment Effect on Change in A1C with Multiple Imputation; Mean Difference (Final Values) = 0.1, 97.5% CI 1-sided [upper limit 0.3]

16. Secondary Outcome: MDI Cohort: Time in Hypoglycemic Range During Night for All Subjects
Description: MDI Cohort: Time with SG below 70 mg/dL (3.9mmol/L) during Night for all subjects
Time Frame: 6 months study period
Population: Study period: 248 subjects in MDI cohort. 206 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | MDI Cohort: Treatment Arm | MDI Cohort: Control Arm
Number analyzed (Participants) | 113 | 93
Percentage of Time | 1.9 (2.6) | 9.2 (14.1)
Statistical Analysis 1: Comparison: MDI Cohort: Treatment Arm vs MDI Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Hypoglycemic Range (%) during Night; Mean Difference (Final Values) = -7.3, 97.5% CI 1-sided [upper limit -4.7]

17. Secondary Outcome: MDI Cohort: Time in Target Range 70mg/dL (3.9mmol/L) - 180 mg/dL (10.0mmol/L) During Night for All Subjects
Description: MDI Cohort: Time in target range measures the time with SG in target range 70mg/dL (3.9mmol/L) - 180 mg/dL (10.0mmol/L) during Night for all subjects
Time Frame: 6 months study period
Population: Study period: 248 subjects in MDI cohort. 206 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | MDI Cohort: Treatment Arm | MDI Cohort: Control Arm
Number analyzed (Participants) | 113 | 93
Percentage of Time | 75.9 (13.6) | 60.0 (21.0)
Statistical Analysis 1: Comparison: MDI Cohort: Treatment Arm vs MDI Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Target Range (%) during Night; Mean Difference (Final Values) = 15.9, 97.5% CI 1-sided [lower limit 11.1]

18. Secondary Outcome: MDI Cohort: Time in Target Range 70mg/dL (3.9mmol/L) - 180 mg/dL (10.0mmol/L) During Day and Night for All Subjects
Description: MDI Cohort: Time in target range measures the time with SG in target range 70mg/dL (3.9mmol/L) - 180 mg/dL (10.0mmol/L) during Day and Night for all subjects
Time Frame: 6 months study period
Population: Study period: 248 subjects in MDI cohort. 208 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | MDI Cohort: Treatment Arm | MDI Cohort: Control Arm
Number analyzed (Participants) | 115 | 93
Percentage of Time | 70.6 (11.3) | 57.0 (15.6)
Statistical Analysis 1: Comparison: MDI Cohort: Treatment Arm vs MDI Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Target Range (%); Mean Difference (Final Values) = 13.6, 97.5% CI 1-sided [lower limit 9.9]

19. Secondary Outcome: MDI Cohort: Time in Hypoglycemic Range During Day and Night for All Subjects
Description: MDI Cohort: Time with SG below 70 mg/dL (3.9mmol/L) during Day and Night for all subjects
Time Frame: 6 months study period
Population: Study period: 248 subjects in MDI cohort. 208 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | MDI Cohort: Treatment Arm | MDI Cohort: Control Arm
Number analyzed (Participants) | 115 | 93
Percentage of Time | 2.4 (2.3) | 6.7 (6.0)
Statistical Analysis 1: Comparison: MDI Cohort: Treatment Arm vs MDI Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Hypoglycemic Range (%); Mean Difference (Final Values) = -4.3, 97.5% CI 1-sided [upper limit -3.1]

20. Secondary Outcome: MDI Cohort: Change in A1C for All Subjects
Description: MDI Cohort: Change in A1C from baseline to the end of the six-month treatment period, defined as A1C measured at the six-month treatment visit minus A1C measured at the randomization visit for all subjects
Time Frame: Baseline and end of 6-month study period
Population: Study period: 248 subjects in MDI cohort. 224 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | MDI Cohort: Treatment Arm | MDI Cohort: Control Arm
Number analyzed (Participants) | 115 | 109
Percentage of HbA1c | -0.6 (1.1) | -0.3 (0.8)
Statistical Analysis 1: Comparison: MDI Cohort: Treatment Arm vs MDI Cohort: Control Arm; Test type: Superiority — Treatment Effect on Change in A1C with Multiple Imputation; Mean Difference (Final Values) = -0.2, 97.5% CI 1-sided [upper limit 0.0]

21. Secondary Outcome: SAP Cohort: Baseline A1C > 8%: Time in Hypoglycemic Range
Description: SAP Cohort: Time with sensor glucose (SG) below 70 mg/dL (3.9mmol/L) during the six-month study period, for subjects with baseline A1c > 8%
Time Frame: 6 months study period
Population: Study period: 324 subjects in SAP cohort. 106 subjects have available measurements in the A1C > 8% group.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | SAP Cohort: Treatment Arm | SAP Cohort: Control Arm
Number analyzed (Participants) | 53 | 53
Percentage of Time | 2.5 (1.9) | 2.8 (3.0)
Statistical Analysis 1: Comparison: SAP Cohort: Treatment Arm vs SAP Cohort: Control Arm; Test type: Non-Inferiority — Non-inferiority margin: 2%. Treatment Effect on Time in Hypoglycemic Range (%) with Multiple Imputation; Mean Difference (Final Values) = -0.3, 97.5% CI 1-sided [upper limit 0.7]

22. Secondary Outcome: SAP Cohort: Baseline A1C ≤ 8%: Change in A1C (∆A1C)
Description: SAP Cohort: Change in A1C from baseline to the end of the six-month treatment period, defined as A1C measured at the six-month treatment visit minus A1C measured at the randomization visit, for subjects with baseline A1c ≤ 8%
Time Frame: Baseline and end of 6-month study period
Population: Study period: 324 subjects in SAP cohort. 184 subjects have available measurements in the baseline A1c ≤ 8% group.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | SAP Cohort: Treatment Arm | SAP Cohort: Control Arm
Number analyzed (Participants) | 92 | 92
Percentage of HbA1c | 0.0 (0.5) | 0.1 (0.5)
Statistical Analysis 1: Comparison: SAP Cohort: Treatment Arm vs SAP Cohort: Control Arm; Test type: Non-Inferiority — Non-inferiority margin: 0.4%. Treatment Effect on Change in A1C with Multiple Imputation; Mean Difference (Final Values) = 0.0, 97.5% CI 1-sided [upper limit 0.1]

23. Secondary Outcome: SAP Cohort: Time in Hypoglycemic Range During Night for All Subjects
Description: SAP Cohort: Time with SG below 70 mg/dL (3.9mmol/L) during Night for all subjects
Time Frame: 6 months study period
Population: Study period: 324 subjects in SAP cohort. 283 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | SAP Cohort: Treatment Arm | SAP Cohort: Control Arm
Number analyzed (Participants) | 142 | 141
Percentage of Time | 2.5 (3.4) | 3.2 (4.4)
Statistical Analysis 1: Comparison: SAP Cohort: Treatment Arm vs SAP Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Hypoglycemic Range (%) during Night; Mean Difference (Final Values) = -0.7, 97.5% CI 1-sided [upper limit 0.2]

24. Secondary Outcome: SAP Cohort: Time in Target Range 70mg/dL (3.9mmol/L) - 180 mg/dL (10.0mmol/L) During Night for All Subjects
Description: SAP Cohort: Time in target range measures the time with SG in target range 70mg/dL (3.9mmol/L) - 180 mg/dL (10.0mmol/L) during Night for all subjects
Time Frame: 6 months study period
Population: Study period: 324 subjects in SAP cohort. 283 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | SAP Cohort: Treatment Arm | SAP Cohort: Control Arm
Number analyzed (Participants) | 142 | 141
Percentage of Time | 73.2 (15.4) | 61.0 (18.4)
Statistical Analysis 1: Comparison: SAP Cohort: Treatment Arm vs SAP Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Target Range (%) during Night; Mean Difference (Final Values) = 12.2, 97.5% CI 1-sided [lower limit 8.3]

25. Secondary Outcome: SAP Cohort: Time in Target Range 70mg/dL (3.9mmol/L) - 180 mg/dL (10.0mmol/L) During Day and Night for All Subjects
Description: SAP Cohort: Time in target range measures the time with SG in target range 70mg/dL (3.9mmol/L) - 180 mg/dL (10.0mmol/L) during Day and Night for all subjects
Time Frame: 6 months study period
Population: Study period: 324 subjects in SAP cohort. 283 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | SAP Cohort: Treatment Arm | SAP Cohort: Control Arm
Number analyzed (Participants) | 142 | 141
Percentage of Time | 65.7 (12.4) | 59.4 (14.0)
Statistical Analysis 1: Comparison: SAP Cohort: Treatment Arm vs SAP Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Target Range (%); Mean Difference (Final Values) = 6.3, 97.5% CI 1-sided [lower limit 3.3]

26. Secondary Outcome: SAP Cohort: Time in Hypoglycemic Range During Day and Night for All Subjects
Description: SAP Cohort: Time with SG below 70 mg/dL (3.9mmol/L) during Day and Night for all subjects
Time Frame: 6 months study period
Population: Study period: 324 subjects in SAP cohort. 283 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | SAP Cohort: Treatment Arm | SAP Cohort: Control Arm
Number analyzed (Participants) | 142 | 141
Percentage of Time | 2.5 (2.2) | 3.3 (3.0)
Statistical Analysis 1: Comparison: SAP Cohort: Treatment Arm vs SAP Cohort: Control Arm; Test type: Superiority — Test of Treatment Effect on Time in Hypoglycemic Range (%); Mean Difference (Final Values) = -0.8, 97.5% CI 1-sided [upper limit -0.1]

27. Secondary Outcome: SAP Cohort: Change in A1C for All Subjects
Description: SAP Cohort: Change in A1C from baseline to the end of the six-month treatment period, defined as A1C measured at the six-month treatment visit minus A1C measured at the randomization visit for all subjects
Time Frame: Baseline and end of 6-month study period
Population: Study period: 324 subjects in SAP cohort. 292 subjects have available measurements.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | SAP Cohort: Treatment Arm | SAP Cohort: Control Arm
Number analyzed (Participants) | 146 | 146
Percentage of HbA1c | -0.2 (0.7) | -0.2 (0.8)
Statistical Analysis 1: Comparison: SAP Cohort: Treatment Arm vs SAP Cohort: Control Arm; Test type: Superiority — Treatment Effect on Change in A1C with Multiple Imputation; Mean Difference (Final Values) = 0.0, 97.5% CI 1-sided [upper limit 0.1]

ADVERSE EVENTS:
Time Frame: 6 months of Study Period, 6 months of Continuation Period
Groups:
- CSII Cohort: Treatment Arm Study Period; MDI Cohort: Treatment Arm Study Period; SAP Cohort: Treatment Arm Study Period: In the study period, subjects started using the MiniMed system (i.e., using Auto Mode).
- CSII Cohort: Control Arm Study Period: In the study period, subjects used the MiniMed pump without CGM.
- MDI Cohort: Control Arm Study Period: In the study period, subjects continued to use MDI.
- SAP Cohort: Control Arm Study Period: In the study period, subjects continued to use SAP therapy using the MiniMed system (SAP without Low Management Suspend on Low, Low Management Suspend before low or Auto Mode).
- All Patients: Continuation Period: In the continuation period, all subjects were using the Hybrid Closed Loop system.
Arm/Group | CSII Cohort: Treatment Arm Study Period | CSII Cohort: Control Arm Study Period | MDI Cohort: Treatment Arm Study Period | MDI Cohort: Control Arm Study Period | SAP Cohort: Treatment Arm Study Period | SAP Cohort: Control Arm Study Period | All Patients: Continuation Period
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/148 | 0/126 | 0/122 | 0/164 | 0/160 | 0/796
Serious Adverse Events (participants affected / at risk) | 1/150 | 4/148 | 3/126 | 2/122 | 4/164 | 6/160 | 26/796
Other Adverse Events (participants affected / at risk) | 80/150 | 86/148 | 72/126 | 77/122 | 94/164 | 101/160 | 395/796
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSII Cohort: Treatment Arm Study Period (N=150) | CSII Cohort: Control Arm Study Period (N=148) | MDI Cohort: Treatment Arm Study Period (N=126) | MDI Cohort: Control Arm Study Period (N=122) | SAP Cohort: Treatment Arm Study Period (N=164) | SAP Cohort: Control Arm Study Period (N=160) | All Patients: Continuation Period (N=796)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSII Cohort: Treatment Arm Study Period (N=150) | CSII Cohort: Control Arm Study Period (N=148) | MDI Cohort: Treatment Arm Study Period (N=126) | MDI Cohort: Control Arm Study Period (N=122) | SAP Cohort: Treatment Arm Study Period (N=164) | SAP Cohort: Control Arm Study Period (N=160) | All Patients: Continuation Period (N=796)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acetonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alveolar osteitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 7 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Artificial crown procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Astigmatism (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 5 (5)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biopsy skin (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood calcium abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood ketone body increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 10 (10)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Calcinosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac stress test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Catheter site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Conjunctival cyst (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 3 (3) | 2 (2) | 5 (7) | 3 (3) | 7 (7)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cystoid macular oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Degenerative bone disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 6 (6)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 8 (8)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Ear lobe infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Essential tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye allergy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye ulcer (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body in reproductive tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 5 (5) | 0 (0) | 3 (4) | 6 (6) | 3 (3) | 16 (20)
Gastroenteritis norovirus (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 10 (10) | 4 (4) | 9 (9)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorder (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival hypertrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival recession (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gluten sensitivity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 3 (3) | 7 (7)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Herpes zoster cutaneous disseminated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hunger (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyalosis asteroid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (13) | 24 (40) | 17 (22) | 3 (3) | 20 (25) | 24 (37) | 70 (97)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 10 (10)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 3 (4) | 2 (2) | 3 (3) | 3 (4) | 4 (4) | 10 (10)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Infusion site abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Infusion site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intersection syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-uterine contraceptive device insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Investigation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lenticular opacities (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (4) | 4 (4)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Mallet finger (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site bruise (General disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Medical device site dermatitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site dryness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site erosion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Medical device site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Medical device site haemorrhage (General disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Medical device site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Medical device site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site injury (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site irritation (General disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Medical device site laceration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Medical device site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Medical device site rash (General disorders) | 1 (1) | 0 (0) | 2 (4) | 2 (2) | 2 (2) | 3 (3) | 7 (7)
Medical device site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 2 (2) | 5 (6)
Medical device site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Medical device site vesicles (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meibomian gland dysfunction (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Mite allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 6 (6)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 9 (11) | 10 (13) | 7 (7) | 10 (10) | 9 (11) | 11 (13) | 52 (56)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-proliferative retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Norovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 6 (6)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 6 (7)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perianal cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 8 (9)
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pinguecula (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Posterior capsule opacification (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Psychological factor affecting medical condition (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 4 (5) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (4) | 3 (4) | 3 (3) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinopathy proliferative (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sever's disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 15 (15)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 5 (5)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Social anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal segmental dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tendon sheath incision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid disorder (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Tractional retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulnocarpal abutment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Infections and infestations) | 6 (7) | 6 (6) | 4 (5) | 10 (10) | 6 (6) | 10 (11) | 35 (37)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (6) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 2 (2) | 16 (19)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 3 (4) | 1 (1) | 5 (6) | 2 (2) | 2 (2) | 2 (2) | 11 (13)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 8 (9) | 1 (1) | 3 (3) | 2 (2) | 10 (11)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees not to publish until 12 months from trial completion or until sponsor publishes multi-center results, whichever occurs first. In either case, sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period more than 60 days but less than or equal to 180 days from the date that the communication is submitted to sponsor for review. Sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT02748018/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT02748018/SAP_001.pdf